CLINICAL TRIAL: NCT02905162
Title: Z 31601 - Understanding Longitudinal Clinical Outcomes and Post-release Retention in Care Among HIV-infected Prisoners in Lusaka, Zambia
Brief Title: Understanding Longitudinal Clinical Outcomes and Post-release Retention in Care Among HIV-infected Prisoners in Lusaka, Zambia
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Other Study IDs: 16-0276; 1K01TW010272-01 (NIH)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: HIV; Alcohol Use Disorders
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV positive individuals incarcerated at Lusaka Central Prison: Cohort of individuals scheduled for release within 30 days will be followed for 6 months post release
  Interventions: Other: Transitional HIV care for prison releasees

INTERVENTIONS:
Other: Transitional HIV care for prison releasees — Transitional HIV care program for releasees

SUMMARY:
To inform the design of a future transitional HIV care intervention for releasees, the study proposes to prospectively assess clinical outcomes for HIV-infected prisoners after release; explore factors from health behavior theory that are associated with post-release retention in care, with a special focus on Alcohol Use Disorders (AUDs); and conduct formative research to determine releasee and stakeholder knowledge, attitudes, and preferences surrounding transitional care interventions.

DETAILED DESCRIPTION:
The study will enrol approximately 552 releasees from Lusaka Central Facility, Mwembeshi Correctional Facility, Kamwala Remand Centre, and Chainama Correctional Facility and Kabwe Correctional Complex. HIV care retention, mortality and changes in CD4 count and HIV-1 viral load at 6 month post-release information will be obtained from the SmartCare database.

Validated psychometric instruments will be used to assess AUD prevalence and alcohol use severity pre-incarceration, at release and about 3 to 6 months post-release. Using mixed-methods, effects of AUDs on retention in care at 3 and/or 6 months post-release will be estimated.

Sub-group analyses among HIV-infected individuals on ART and those enrolled in care but not yet on ART (i.e. pre-ART) will enable assessment of AUD effects on biological markers of HIV disease control and progression.

The Behavioural Model for Vulnerable Populations, and validated psychometric instruments, questionnaires, and in-depth interviews, factors beyond AUDs that may influence post-release retention in HIV care will be evaluated. Finally, preferred and relevant program elements for a future prisoner transitional HIV care pilot will be examined by conducting in-depth interviews with a purposive sample of approximately 26 HIV-infected releasees and leaders from the Zambian government and prominent implementing partner organizations, as well as focus group discussions with frontline prison officers, health workers, and representatives of leading civil society organizations in Zambia.

ELIGIBILITY:
Participant inclusion criteria

* Currently incarcerated a
* Release scheduled or otherwise anticipated within 30 days
* Has documented HIV infection
* Enrolled in the national HIV programme while in prison (i.e. receiving ART, receiving pre- ART care, or otherwise followed by the national HIV programme)
* If on treatment, has been receiving ART for approximately ≥3 months
* Plan to live in Lusaka Urban district after release
* Willing and able to provide locator information, including a reachable telephone number
* Willing and able to provide informed consent in Nyanja, Bemba, or English, including agreeing to be contacted by study staff after release and be followed for 6 mo. after discharge.

Participant exclusion criteria

* < 18 years of age
* Residing outside Lusaka district before incarceration
* Remandees awaiting trial who have been detained for less than 180 days
* Offenders being held at Lusaka Central Prison while awaiting appeal of a capital offence (e.g.murder or rape) or who have had their current sentence extended for violent behaviour during their period of incarceration.

Focus Group Discussion Participant Eligibility:

* Must be 18 years of age or older
* Working in Corrections or health as a corrections health manager, facility manager, or other corrections officers OR MOH clinician, nurse, physician or peer health educator OR member of a civil society or implementing partner organization working on corrections health.
* Able to provide verbal informed consent in English

Key Stakeholder in-depth Interview Participant eligibility criteria:

* Must be 18 years of age or older
* Involved in corrections and/or health policy making in Zambia
* Able to provide verbal informed consent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected inmates who are scheduled for release, including those not yet qualifying for ART (pre-ART), those on ART based on Zambian Treatment Guidelines, and those who qualify for ART but who have refused to start treatment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Number of prison releasees retained in care | 6 months post release
  number of participants known to be alive with at least one clinical encounter in the national HIV program documented

SECONDARY OUTCOMES:
Number virologically suppressed | 6 months post release (release for ART-treated releasees)
Change in CD4 count | 6 months post-release
  for HIV-infected releasees not yet on ART

CONTACTS AND LOCATIONS:
Overall Officials: Michael Herce, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia